CLINICAL TRIAL: NCT00627549
Title: The Use of Avaulta Plus for Anterior Repair. A Multicenter Randomised Prospective Controlled Study
Brief Title: Avaulta Versus Anterior Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Other Study IDs: Avaulta 17431
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Vaginal Prolapse
Keywords: cystocele, anterior repair, mesh
MeSH Terms: conditions — Uterine Prolapse; Cystocele

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Avaulta (surgical procedure using a mesh implant)
- 2 (Active Comparator)
  Interventions: Procedure: Conventional surgery (anterior repair)

INTERVENTIONS:
Procedure: Avaulta (surgical procedure using a mesh implant) — The use of Avaulta
  Arms: 1
Procedure: Conventional surgery (anterior repair) — Anterior repair surgery
  Arms: 2

SUMMARY:
Summary:

Vaginal prolapse is a well-known disease and is observed in approximately 11% of all postmenopausal women and tending to increase with age. Consequently, many surgical procedures have been developed in order to ensure sufficient support for the bladder, rectum or vaginal vault depending on the site of the defect. However, many procedures are associated with a high recurrence rate up to 40 % even within one to two years after the surgical procedure.

Due to the high recurrence rate new methods include the use of mesh, either biologically or synthetic. The latter is a permanent implant and therefore theoretically may result in a long-lasting anatomically correct position of the prolapse.

Although the recurrence rate may be lower using a mesh such surgical procedures may be associated with adverse events such as erosions of the vaginal mucosa. Others have observed shrinkage of the vaginal mucosa. However, in these studies large prolene mesh have been used. In contrast the recurrence rate is lowered up to 25%.

The above-mentioned advantage of synthetic mesh is however, mostly based on few non-randomised studies. We therefore find it of importance to evaluate whether a surgical procedure using a mesh implant is superior to conventional surgical techniques. The present study is a clinical controlled study where patients with anterior vaginal prolapse are randomised to either a mesh technique or a standard anterior procedure.

The present study includes only two more visits at the outpatient clinic after the surgical procedure. Furthermore the patients have to fulfil questionnaires regarding urinary and faecal leakage and sexual habits.

Any participation in the study is totally voluntary and the patient may at any time withdraw herself. In any case the patient will receive our standard treatment.

The study is performed in all the Scandinavian countries.

ELIGIBILITY:
Inclusion Criteria:

* Women aged > 55 yr
* Women with anterior vaginal wall prolapse stage >2 according to POP-Q classification
* Good understanding the language in word and writing

Exclusion Criteria:

* A history of previous major pelvic surgery with the exception of a hysterectomy for reasons other than genital prolapse
* Patients with previous vaginal surgery because of defects in the anterior of posterior compartments
* Previous hysterectomy because of vaginal prolapse
* Patients with prolapse of uterus or an enterocele > stage 2
* Patients with previous TVT performed through the obturator membrane
* History of genital or abdominal cancer
* Patients treated with corticosteroids
* Not able to understand the study protocol (language problems, cognitive dysfunction etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Does Avaulta Plus reduce the recurrence rate defined as a POP-Q Aa <-2 cm at follow-up after 1 yr. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Roskilde University Hospital, Roskilde, Denmark

REFERENCES:
- [Derived] Rudnicki M, Laurikainen E, Pogosean R, Kinne I, Jakobsson U, Teleman P. A 3-year follow-up after anterior colporrhaphy compared with collagen-coated transvaginal mesh for anterior vaginal wall prolapse: a randomised controlled trial. BJOG. 2016 Jan;123(1):136-42. doi: 10.1111/1471-0528.13628. Epub 2015 Sep 30. PMID 26420345
- [Derived] Teleman P, Laurikainen E, Kinne I, Pogosean R, Jakobsson U, Rudnicki M. Relationship between the Pelvic Organ Prolapse Quantification system (POP-Q), the Pelvic Floor Impact Questionnaire (PFIQ-7), and the Pelvic Floor Distress Inventory (PFDI-20) before and after anterior vaginal wall prolapse surgery. Int Urogynecol J. 2015 Feb;26(2):195-200. doi: 10.1007/s00192-014-2434-6. Epub 2014 May 28. PMID 24866279
- [Derived] Rudnicki M, Laurikainen E, Pogosean R, Kinne I, Jakobsson U, Teleman P. Anterior colporrhaphy compared with collagen-coated transvaginal mesh for anterior vaginal wall prolapse: a randomised controlled trial. BJOG. 2014 Jan;121(1):102-10; discussion 110-1. doi: 10.1111/1471-0528.12454. Epub 2013 Oct 1. PMID 24118844